CLINICAL TRIAL: NCT01418261
Title: Renal Denervation in Patients With Uncontrolled Hypertension (SYMPLICITY HTN-3)
Brief Title: SYMPLICITY HTN-3 Renal Denervation in Patients With Uncontrolled Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP125
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Uncontrolled Hypertension
Keywords: uncontrolled hypertension; renal denervation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation (Experimental): Subjects are treated with the renal denervation procedure after randomization and maintained baseline anti-hypertensive medications
  Interventions: Device: Renal denervation (Symplicity Catheter System); Diagnostic Test: Renal angiogram
- Control group (Sham Comparator): Subjects go through renal angiogram and Subjects maintained baseline anti-hypertensive medications
  Interventions: Diagnostic Test: Renal angiogram

INTERVENTIONS:
Device: Renal denervation (Symplicity Catheter System)
  Arms: Renal Denervation
Diagnostic Test: Renal angiogram

SUMMARY:
The Symplicity HTN-3 study is a, multi-center, prospective, single-blind, randomized, controlled study of the safety and effectiveness of renal denervation in subjects with uncontrolled hypertension. Bilateral renal denervation will be performed using the Symplicity Catheter - a percutaneous system that delivers radiofrequency (RF)energy through the luminal surface of the renal artery.

DETAILED DESCRIPTION:
The Symplicity HTN-3 study is a, multi-center, prospective, single-blind, randomized, controlled study of the safety and effectiveness of renal denervation in subjects with uncontrolled hypertension. Bilateral renal denervation will be performed using the Symplicity Catheter - a percutaneous system that delivers radiofrequency (RF)energy through the luminal surface of the renal artery.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥ 18 and ≤ 80 years old at time of randomization.
* Individual is receiving a stable medication regimen including full tolerated doses of 3 or more anti-hypertensive medications of different classes, of which one must be a diuretic (with no changes for a minimum of 2 weeks prior to screening) that is expected to be maintained without changes for at least 6 months.
* Individual has an office systolic blood pressure (SBP) of ≥ 160 mmHg based on an average of 3 blood pressure readings measured at both an initial screening visit and a confirmatory screening visit

Exclusion Criteria:

* Individual has an estimated glomerular filtration rate (eGFR) of < 45 mL/min/1.73 m2
* Individual has an Ambulatory Blood Pressure Monitoring (ABPM) 24 hour average SBP < 135 mmHg
* Individual has type 1 diabetes mellitus
* Individual requires chronic oxygen support or mechanical ventilation (e.g., tracheostomy, CPAP, BiPAP) other than nocturnal respiratory support for sleep apnea.
* Individual has primary pulmonary hypertension.
* Individual is pregnant, nursing or planning to be pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Office Systolic Blood Pressure | Baseline to 6 months post-randomization
  Primary Effectiveness Outcome Measure

SECONDARY OUTCOMES:
Change in average 24-hour Systolic Blood Pressure by ambulatory blood pressure monitoring | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, MD, Principal Investigator — Professor of Medicine, Hypertension Center Director University of Chicago Medical Center; Deepak L Bhatt, MD, MPH, Principal Investigator — VA Boston Healthcare System Department of Cardiology
Locations (79):
- United States (79):
  - Cardiology, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scripps Clinic/Scripps Green Hospital, La Jolla, California
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - St. Joseph Hospital, Orange, California
  - San Diego Cardiac Center, San Diego, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Shands / University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - Baptist Cardiac &Vascular Institute, Baptist Health Systems, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Midwest Heart Foundation, Oakbrook Terrace, Illinois
  - Prairie Heart Institute, Springfield, Illinois
  - Iowa Heart Center Research, Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital - Detroit Medical Center, Detroit, Michigan
  - St Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Providence Hospital, Southfield, Michigan
  - Michigan Heart, St. Joseph Mercy Health System, Ypsilanti, Michigan
  - Abbott Northwestern/Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Mary's Mayo Clinic, Rochester, Minnesota
  - Hattiesburg Clinic, P.A, Hattiesburg, Mississippi
  - Saint Luke's Hospital of Kansas City/Mid America Heart Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Medical Center-Manhattan, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Stony Brook University Hospital and Medical Center, Stony Brook, New York
  - University of North Carolina Heart and Vascular, Chapel Hill, North Carolina
  - Carolinas Healthcare (SHVI)-Clinical Research, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Thomas Jefferson University Hospitals, Inc, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Vascular Disease Research Center at Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Inc., Memphis, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Austin Heart PLLC / Heart Hospital of Austin, Austin, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Soltero Cardiovascular Research Center - Baylor Jack and Jane Hamilton Heart & Vascular Hospital, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt DL, Vaduganathan M, Kandzari DE, Leon MB, Rocha-Singh K, Townsend RR, Katzen BT, Oparil S, Brar S, DeBruin V, Fahy M, Bakris GL; SYMPLICITY HTN-3 Steering Committee Investigators. Long-term outcomes after catheter-based renal artery denervation for resistant hypertension: final follow-up of the randomised SYMPLICITY HTN-3 Trial. Lancet. 2022 Oct 22;400(10361):1405-1416. doi: 10.1016/S0140-6736(22)01787-1. Epub 2022 Sep 18. PMID 36130612
- [Derived] Mahfoud F, Bakris G, Bhatt DL, Esler M, Ewen S, Fahy M, Kandzari D, Kario K, Mancia G, Weber M, Bohm M. Reduced blood pressure-lowering effect of catheter-based renal denervation in patients with isolated systolic hypertension: data from SYMPLICITY HTN-3 and the Global SYMPLICITY Registry. Eur Heart J. 2017 Jan 7;38(2):93-100. doi: 10.1093/eurheartj/ehw325. PMID 28158510
- [Derived] Pocock SJ, Bakris G, Bhatt DL, Brar S, Fahy M, Gersh BJ. Regression to the Mean in SYMPLICITY HTN-3: Implications for Design and Reporting of Future Trials. J Am Coll Cardiol. 2016 Nov 1;68(18):2016-2025. doi: 10.1016/j.jacc.2016.07.775. PMID 27788856
- [Derived] Kario K, Bhatt DL, Brar S, Cohen SA, Fahy M, Bakris GL. Effect of Catheter-Based Renal Denervation on Morning and Nocturnal Blood Pressure: Insights From SYMPLICITY HTN-3 and SYMPLICITY HTN-Japan. Hypertension. 2015 Dec;66(6):1130-7. doi: 10.1161/HYPERTENSIONAHA.115.06260. Epub 2015 Oct 5. PMID 26558819
- [Derived] Bakris GL, Townsend RR, Flack JM, Brar S, Cohen SA, D'Agostino R, Kandzari DE, Katzen BT, Leon MB, Mauri L, Negoita M, O'Neill WW, Oparil S, Rocha-Singh K, Bhatt DL; SYMPLICITY HTN-3 Investigators. 12-month blood pressure results of catheter-based renal artery denervation for resistant hypertension: the SYMPLICITY HTN-3 trial. J Am Coll Cardiol. 2015 Apr 7;65(13):1314-1321. doi: 10.1016/j.jacc.2015.01.037. PMID 25835443
- [Derived] Kandzari DE, Bhatt DL, Brar S, Devireddy CM, Esler M, Fahy M, Flack JM, Katzen BT, Lea J, Lee DP, Leon MB, Ma A, Massaro J, Mauri L, Oparil S, O'Neill WW, Patel MR, Rocha-Singh K, Sobotka PA, Svetkey L, Townsend RR, Bakris GL. Predictors of blood pressure response in the SYMPLICITY HTN-3 trial. Eur Heart J. 2015 Jan 21;36(4):219-27. doi: 10.1093/eurheartj/ehu441. Epub 2014 Nov 16. PMID 25400162
- [Derived] Bakris GL, Townsend RR, Liu M, Cohen SA, D'Agostino R, Flack JM, Kandzari DE, Katzen BT, Leon MB, Mauri L, Negoita M, O'Neill WW, Oparil S, Rocha-Singh K, Bhatt DL; SYMPLICITY HTN-3 Investigators. Impact of renal denervation on 24-hour ambulatory blood pressure: results from SYMPLICITY HTN-3. J Am Coll Cardiol. 2014 Sep 16;64(11):1071-8. doi: 10.1016/j.jacc.2014.05.012. Epub 2014 May 20. PMID 24858423
- [Derived] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939